CLINICAL TRIAL: NCT01009385
Title: Cervical Epidural Pressure Measurement: Comparison in the Prone and Sitting Positions
Brief Title: Cervical Epidural Pressure Measurement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Jeeyoun Moon/Instructor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: snu23802
Record Dates: First submitted 2009-11-04; First posted 2009-11-06 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Head Pain; Neck Pain; Upper Extremity Pain
Keywords: cervical; epidural; epidural pressure; monitoring
MeSH Terms: conditions — Headache; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prone position (Active Comparator)
  Interventions: Procedure: cervical epidural steroid injection; Procedure: epidural pressure measurement
- sitting position (Active Comparator)
  Interventions: Procedure: cervical epidural steroid injection; Procedure: epidural pressure measurement

INTERVENTIONS:
Procedure: cervical epidural steroid injection — * After aseptic preparation and skin infiltration with 1% lidocaine
  * 20-gauge Tuohy needle (Tae-Chang Industrial Co., Kongju, Korea) was inserted in the midline at the C6 - C7 level
  * identification of the epidural space confirmed by injection of contrast medium under fluoroscope
  * injection of 5 mL of solution containing 10 mg of triamcinolone acetonide suspension and 1.5 mL of 0.75% levobupivacaine hydrochloride, and 3.5 mL of physiologic saline (0.9% NaCl).
  * Post-procedure, patients were observed for any adverse effects and followed with a neurological examination
  Other Names: cervical interlaminar epidural injection
Procedure: epidural pressure measurement — * The stylet within the Tuohy needle is removed when the needle was placed in C6-7 ligamentum flavum under fluoroscopic true lateral view.
  * Identification of the epidural space and measurement of EP was performed with a closed measurement system.
  Other Names: a closed pressure measurement system

SUMMARY:
Cervical epidural steroid injections

* The hanging drop (HD) technique is commonly used for identifying the cervical epidural space.
* The hanging drop (HD) technique is using the negative pressure in the epidural space.
* The subject of debate whether the epidural space exhibits negative pressure.
* In a previous study, EP might be influenced by body position
* No report or peer-reviewed literature to demonstrate the cervical epidural pressure (CEP) now.

The hypothesis of this study

* There is a difference in the cervical epidural pressure between in the prone and sitting positions
* To evaluate this hypothesis, CEPs in the prone and sitting groups were measured and compared in the two groups.
* Using a closed pressure measurement system
* Under fluoroscopic guidance.

DETAILED DESCRIPTION:
Cervical epidural steroid injections (CESIs)

* For the conservative management of head, neck, and upper extremity pain
* Important to identify the epidural space for minimizing the chance of a dural puncture injection
* Dural puncture injection makes CESIs prone to rare but catastrophic complication like permanent spinal cord injury

The hanging drop (HD) technique

* Commonly used for identifying the cervical epidural space
* Using the negative pressure in the epidural space
* The subject of debate whether the epidural space exhibits negative pressure

In previous studies using a closed pressure measurement systems

* The epidural pressure (EP) was commonly positive at the thoracic level in the lateral decubitus position.
* EP was consistently negative only in the sitting position.
* EP might be influenced by body position.
* The patient should be sitting for using the HD technique.

No report or peer-reviewed literature to demonstrate the cervical epidural pressure (CEP) now.

The hypothesis of this study

* There is a difference in the cervical epidural pressure between in the prone and sitting positions
* To evaluate this hypothesis, CEPs in the prone and sitting groups were measured and compared in the two groups.
* Using a closed pressure measurement system
* Under fluoroscopic guidance.

ELIGIBILITY:
Inclusion Criteria:

* cervical radicular pain caused by herniated nucleus pulpous and spinal stenosis
* other conditions including herpes zoster-associated pain and sprain.

Exclusion Criteria:

* contraindications for CESIs, such as coagulopathy, patient refusal or infection at the proposed insertion site
* previous cervical spinal surgery
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
cervical epidural pressure | on interventional procedure (cervical epidural steroid injetion)

SECONDARY OUTCOMES:
the angle of the neck flexion | on interventional procedure (cervical epidural steroid injection)

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyoun Moon, Principal Investigator — Department of Anesthesiology and Pain Medicine, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Kŭmi, Kyonggi-do, South Korea

REFERENCES:
- [Derived] Joo Y, Moon JY, Kim YC, Lee SC, Kim HY, Park SY. A pressure comparison between midline and paramedian approaches to the cervical epidural space. Pain Physician. 2014 Mar-Apr;17(2):155-62. PMID 24658476
- [Derived] Moon JY, Lee PB, Nahm FS, Kim YC, Choi JB. Cervical epidural pressure measurement: comparison in the prone and sitting positions. Anesthesiology. 2010 Sep;113(3):666-71. doi: 10.1097/ALN.0b013e3181e898e8. PMID 20693880